CLINICAL TRIAL: NCT00681070
Title: Cosmetic Outcomes of Absorbable Versus Non-absorbable Sutures in Pediatric Facial Lacerations, Part 2
Brief Title: Cosmetic Outcomes of Absorbable Versus Non-absorbable Sutures in Pediatric Facial Lacerations
Acronym: Catgut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11020; 11020-2
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Lacerations; Wounds
Keywords: laceration; wound management; absorbable sutures; cosmetic outcomes
MeSH Terms: conditions — Lacerations; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm1: Non-absorbable sutures (Active Comparator): use of non-absorbable sutures in facial laceration in this arm
  Interventions: Other: Arm 1: non-absorbable sutures
- Arm 2: Absorbable sutures (Active Comparator): use of absorbable sutures in this arm
  Interventions: Other: Arm 2: Absorbable sutures

INTERVENTIONS:
Other: Arm 2: Absorbable sutures — use of absorbable catgut sutures in pediatric facial lacerations
  Other Names: fast-absorbing catgut 5-0 by Johnson and Johnson
  Arms: Arm 2: Absorbable sutures
Other: Arm 1: non-absorbable sutures — Use of non-absorbing sutures
  Arms: Arm1: Non-absorbable sutures

SUMMARY:
Our research hypothesis in this study is that there is no difference in long-term cosmetic outcomes between absorbable sutures and non-absorbable sutures in the repair of pediatric facial lacerations.

DETAILED DESCRIPTION:
The standard method of repair for facial lacerations is to close such wounds with non-absorbable sutures. Recently, topical skin adhesives such as n-butyl-2-cyanoacrylate and 2-octyl cyanoacrylate have been used more frequently as these have been shown to be a faster and less painful way to close superficial facial lacerations. However, lacerations that are deeper, gaping or occurring along lines of excessive tension, such as the chin, still need sutures for repair. Non-absorbable sutures have to be taken out at 4-7 days. This involves another physician visit, parental absence from work, and children who need to be taken out of school or daycare for a simple suture removal.

In Part Iof the study, we were able to demonstrate non-inferiority of absorbable sutures to nylon sutures. However, we purposely removed all remaining absorbable sutures on the 5-7 day follow-up visit. In Part II, we will allow the absorbable sutures to dissolve on their own. We will again assess long term cosmetic outcomes, as well parental satisfaction, and short and long-term complication rates at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Clean. minimally contaminated facial lacerations, between 1-5 cms long, less than 8 hours old, not caused by animal bites, not needing plastic surgery repair

Exclusion Criteria:

* Pregnancy
* Bleeding
* Renal
* Endocrine problems
* Dirty wounds
* Irregular wounds

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
cosmetic outcomes | 3 months

SECONDARY OUTCOMES:
infection | 4-6 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Temple University Hospital, Philadelphia, Pennsylvania